CLINICAL TRIAL: NCT06701838
Title: Osilodrostat Therapy and 11C-methionine PET to IMprove Corticotroph Pituitary Adenoma Detection and Localisation in Patients With Cushing's Disease
Brief Title: Osilodrostat Therapy and 11C-methionine PET to Improve Corticotroph Adenoma Detection
Acronym: OPTIMAL
Status: Not yet recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Sponsor
Other Study IDs: 24/EM/0178
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Cushing's Disease; Hypercortisolism; Pituitary Adenoma; Pituitary ACTH Secreting Adenoma
Keywords: Cushing's disease; Osilodrostat; 11C-methionine PET; Corticotroph adenoma
MeSH Terms: conditions — Cushing Syndrome; Pituitary Neoplasms; Pituitary ACTH Hypersecretion; ACTH-Secreting Pituitary Adenoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples, pituitary tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 11C-Methionine PET/CT — After a 3-month period of eucortisolaemia, patients will undergo a second MRI of the pituitary gland and 11C-methionine PET/CT scan with SUVmax ratio analysis of the presumed corticotroph pituitary adenoma.

SUMMARY:
Cushing's disease is a rare condition where the body produces too much of a hormone called cortisol. Cortisol helps with metabolism, the immune system, and managing stress. But too much cortisol can lead to problems like weight gain, high blood pressure, diabetes, and changes in appearance, such as a round face or a hump on the back. People with Cushing's disease often gain weight around their belly and may get stretch marks. They might also feel emotional changes, tiredness, or weakness. This disease is usually caused by a small, non-cancerous growth in the pituitary gland called a 'pituitary adenoma.' The pituitary gland is a small organ at the base of the brain and controls many important functions.

When someone is diagnosed with Cushing's disease, doctors typically use an MRI scan to look for the adenoma in the pituitary gland. If found, the adenoma can often be removed through surgery, which often cures the disease. This is the standard treatment for patients with Cushing's disease. However, MRIs only find the adenoma in about 60% of the time. If surgery isn't possible because the adenoma can't be located, doctors may use medication to lower cortisol levels.

In addition to the MRI, doctors might use a special PET/CT scan to find the adenoma. This PET/CT scan is not available everywhere, so the investigators refer our patients to Cambridge Hospital for this scan, which uses a special dye called 11C-methionine.

The investigators then review the scan with the teams from Imperial and Cambridge. If the PET/CT scan shows where the adenoma is, the patient will be offered surgery. However, finding the adenoma can be challenging because they are often small and hard to distinguish from normal tissue.

If the adenoma isn't visible, the investigators will use medical treatment to lower cortisol. After a period of medical treatment, another MRI scan and PET/CT scan will be done to see if the adenoma has become clearer. This second PET/CT scan would not normally be part of routine clinical care. The investigators will then compare the results of the two scans to see if the special dye is showing a stronger signal, which can help us find the adenoma more accurately and improve the chance of curing Cushing's disease with surgery.

DETAILED DESCRIPTION:
BACKGROUND Cushing's disease is a rare endocrine disorder caused by the overproduction of adrenocorticotropic hormone (ACTH) from a corticotroph pituitary adenoma. It accounts for approximately 15% of all pituitary adenomas and has a female predominance (4:1). Cushing's disease is associated with increased mortality, substantial morbidity, and a notable impact on health-related quality of life. Diagnosis involves a variety of assessments, including demonstration of autonomous ACTH-driven hypercortisolaemia, inferior petrosal sinus sampling to exclude an ectopic source of ACTH production and MRI of the pituitary gland to identify a pathological pituitary adenoma.

Trans-sphenoidal surgical (TSS) resection of a pituitary adenoma remains the primary treatment. However, the surgical cure rate only ranges between 60% and 80% and therefore, repeated pituitary surgery, pituitary radiotherapy, or bilateral adrenalectomy are often required to achieve cure. Pre-operative medical (cortisol-lowering) therapy reduces both morbidity and perioperative complications. Both ketoconazole and metyrapone have been used as cortisol-lowering treatments, but effectiveness can be variable and adverse side effects are often significant necessitating dose reduction.

Osilodrostat, a potent inhibitor of the enzyme 11-beta-hydroxylase has been shown to be highly effective in normalising urinary free cortisol levels and achieving clinical remission in patients with Cushing's disease. The Phase III LINC-3 study investigated the efficacy and safety of osilodrostat in patients with Cushing's disease who were ineligible for pituitary surgery or had previously undergone unsuccessful pituitary surgery. The trial revealed that osilodrostat successfully normalised urinary free cortisol levels in a significant proportion of patients leading to improvements in clinical signs and symptoms of Cushing's disease. Importantly, the study reported a very favourable side effect and safety profile for Osilodrostat.

In Cushing's disease, dedicated pituitary MRI only identifies a suitable surgical target in 60% of cases. Recently, 11C-methionine PET/CT has emerged as a valuable additional tool for the localisation of pituitary lesions not clearly identified with conventional MRI. 11C-methionine is taken up by peptide-secreting cells via the L-type amino acid transporter 1 (LAT1), which is expressed in pituitary tissue, including pituitary adenomas. Functioning pituitary adenomas such as somatotroph adenomas, prolactinomas and, to a lesser extent, corticotroph adenomas, show increased uptake of 11C-methionine compared to normal pituitary tissue, and this can allow accurate localisation of small tumours that are not clearly visualised on anatomical imaging, as well as discriminate between post-surgical tissue re-modelling and residual tumour in patients who have undergone previous unsuccessful surgery.

Treatment with osilodrostat is associated with an increase in circulating ACTH levels, reflecting reduction in adrenal glucocorticoid biosynthesis by osilodrostat with consequent attenuation of negative feedback by cortisol at the level of the hypothalamus and pituitary, but also corticotroph pituitary adenomas, as corticotroph adenomas, albeit autonomously ACTH-producing, appear to retain a degree of feedback regulation. The investigators predict that the lack of negative feedback may lead to an increase in corticotroph tumour activity, thereby improving radiological detection of corticotroph tumours not seen on imaging prior to osilodrostat treatment.

The investigators therefore hypothesise that a period of medical treatment with osilodrostat may enhance the detection and localisation of corticotroph adenomas by using 11C-methionine PET.

RATIONALE FOR CURRENT STUDY Even with the adoption of modern and innovative MR sequences, an important subgroup of corticotroph tumours cannot be readily localised. Whilst the introduction of molecular imaging with 11C-methionine PET/CT can aid detection of a proportion of such occult tumours, we believe that detection could be further enhanced by repeating 11C-methionine PET/CT following a period of medical treatment. The possible increase in tumoral activity during the period of medical treatment would be anticipated to correlate with increased 11C-methionine uptake. A period of treatment with osilodrostat (the most effective cortisol-lowering medical treatment available) prior to surgery and resulting reduced negative feedback due to reduction of excess cortisol levels, might in turn enhance the clarity of both conventional and functional imaging and might aid the identification of previously occult adenomas.

STUDY OBJECTIVES This observational study is to investigate whether the combination of treatment with osilodrostat and 11C-methionine PET/CT may help to identify occult/ equivocal pituitary corticotroph adenomas in patients with Cushing's disease.

• Change in 11C-methionine SUVmax in a presumed corticotroph adenoma through comparison of pre- and post-osilodrostat 11C-methionine PET/CT.

STUDY DESIGN OPTIMAL is a single-arm observational study. The inclusion and exclusion criteria are listed in Section 4, but in brief, the study population will consist of adult patients diagnosed with Cushing's disease according to Endocrine Society Guidelines with no/ an equivocal surgical target on MRI pituitary.

The visit schedule and data collection are detailed in appendix.

STUDY OUTCOME MEASURES Primary outcome • Tumour activity on functional imaging Change in 11C-methionine SUVmax in a corticotroph adenoma through comparison of pre- and post-osilodrostat 11C-methionine PET/CT.

Secondary outcomes

• Radiological tumour appearance Change in MRI appearance of a presumed corticotroph adenoma pre- and post-osilodrostat treatment.

INCLUSION CRTERIA

All participants must meet all of the following inclusion criteria:

* age 18 years and older newly diagnosed with Cushing's disease and no/ an equivocal surgical target on MRI pituitary or
* age 18 years and older and previously undergone pituitary surgery for Cushing's disease and clinical and biochemical evidence of persistent/ recurrent hypercortisolaemia and no/ an equivocal surgical target on MRI pituitary.

EXCLUSION CRITERIA

Potential participants will be ineligible to enter the study if they meet any of the following exclusion criteria:

* Absolute contraindication to osilodrostat therapy and/or 11C methionine PET.
* Pregnancy or unwillingness to use secure contraception for the study duration (female participants only).
* Unable to comply with study visit schedule.

STUDY PROCEDURE A total of 15 patients with confirmed Cushing's disease will be enrolled and undergo baseline assessments including MRI of the pituitary gland and 11C-methionine PET/CT. Patients will start medical therapy with osilodrostat as per our local standard practice and will follow a titration regimen as described in the Phase III LINC-3 study, with the aim to normalise UFC levels for a period of at least 3 months.

Preferably, an osilodrostat titration-based approach will be used and a block-and-replace regimen will be reserved for patients in whom normalisation of cortisol levels cannot safely be achieved with titration of osilodrostat alone. After a 3-month period of eucortisolaemia, patients will undergo a second MRI of the pituitary gland and 11C-methionine PET/CT scan with SUVmax ratio analysis of the presumed corticotroph pituitary adenoma.

Comparison between the first and second 11C-methionine PET/CT will be carried out and a change of >20% in SUVmax constitutes a positive result.

Additionally, this observational study will collect data on biochemical markers of bone health, cardiovascular health, hypercoagulopathy, and quality of life. However, it is important to note that such data are for descriptive purposes only and are being collected as they may be useful as groundwork for a potential larger prospective study in the future.

ELIGIBILITY:
Inclusion Criteria:

All participants must meet all of the following inclusion criteria:

* age 18 years and older newly diagnosed with Cushing's disease and no/ an equivocal surgical target on MRI pituitary or
* age 18 years and older and previously undergone pituitary surgery for Cushing's disease and clinical and biochemical evidence of persistent/ recurrent hypercortisolaemia and no/ an equivocal surgical target on MRI pituitary.

Exclusion Criteria:

Potential participants will be ineligible to enter the study if they meet any of the following exclusion criteria:

* Absolute contraindication to osilodrostat therapy and/or 11C methionine PET.
* Pregnancy or unwillingness to use secure contraception for the study duration (female participants only).
* Unable to comply with study visit schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Following confirmation of eligibility patient's will be discussed at a pre-enrolment MDT before recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-12-03 (Estimated); Primary Completion 2026-07-05 (Estimated); Study Completion 2026-07-05 (Estimated)

PRIMARY OUTCOMES:
Tumour activity on functional imaging | Following 3-month period of eucortisolaemia
  Change in 11C-methionine SUVmax in a corticotroph adenoma through comparison of pre- and post-osilodrostat 11C-methionine PET/CT

SECONDARY OUTCOMES:
Radiological tumour appearance | Following a 3-month period of eucortisolaemia.
  Change in MRI appearance of a presumed corticotroph adenoma pre- and post-osilodrostat treatment.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gillett D, Senanayake R, MacFarlane J, van der Meulen M, Koulouri O, Powlson AS, Crawford R, Gillett B, Bird N, Heard S, Kolias A, Mannion R, Aloj L, Mendichovszky IA, Cheow H, Bashari WA, Gurnell M. Localization of TSH-secreting pituitary adenoma using 11C-methionine image subtraction. EJNMMI Res. 2022 May 7;12(1):26. doi: 10.1186/s13550-022-00899-7. PMID 35524902
- [Background] Bashari WA, van der Meulen M, MacFarlane J, Gillett D, Senanayake R, Serban L, Powlson AS, Brooke AM, Scoffings DJ, Jones J, O'Donovan DG, Tysome J, Santarius T, Donnelly N, Boros I, Aigbirhio F, Jefferies S, Cheow HK, Mendichovszky IA, Kolias AG, Mannion R, Koulouri O, Gurnell M. 11C-methionine PET aids localization of microprolactinomas in patients with intolerance or resistance to dopamine agonist therapy. Pituitary. 2022 Aug;25(4):573-586. doi: 10.1007/s11102-022-01229-9. Epub 2022 May 24. PMID 35608811
- [Background] Bashari WA, Gillett D, MacFarlane J, Powlson AS, Kolias AG, Mannion R, Scoffings DJ, Mendichovszky IA, Jones J, Cheow HK, Koulouri O, Gurnell M. Modern imaging in Cushing's disease. Pituitary. 2022 Oct;25(5):709-712. doi: 10.1007/s11102-022-01236-w. Epub 2022 Jun 6. PMID 35666391
- [Background] Lonser RR, Nieman L, Oldfield EH. Cushing's disease: pathobiology, diagnosis, and management. J Neurosurg. 2017 Feb;126(2):404-417. doi: 10.3171/2016.1.JNS152119. Epub 2016 Apr 22. PMID 27104844
- [Background] Gadelha M, Bex M, Feelders RA, Heaney AP, Auchus RJ, Gilis-Januszewska A, Witek P, Belaya Z, Yu Y, Liao Z, Ku CHC, Carvalho D, Roughton M, Wojna J, Pedroncelli AM, Snyder PJ. Randomized Trial of Osilodrostat for the Treatment of Cushing Disease. J Clin Endocrinol Metab. 2022 Jun 16;107(7):e2882-e2895. doi: 10.1210/clinem/dgac178. PMID 35325149
- [Background] Biller BM, Grossman AB, Stewart PM, Melmed S, Bertagna X, Bertherat J, Buchfelder M, Colao A, Hermus AR, Hofland LJ, Klibanski A, Lacroix A, Lindsay JR, Newell-Price J, Nieman LK, Petersenn S, Sonino N, Stalla GK, Swearingen B, Vance ML, Wass JA, Boscaro M. Treatment of adrenocorticotropin-dependent Cushing's syndrome: a consensus statement. J Clin Endocrinol Metab. 2008 Jul;93(7):2454-62. doi: 10.1210/jc.2007-2734. Epub 2008 Apr 15. PMID 18413427
- [Background] Wang B, Zheng S, Ren J, Zhong Z, Jiang H, Sun Q, Su T, Wang W, Sun Y, Bian L. Reoperation for Recurrent and Persistent Cushing's Disease without Visible MRI Findings. J Clin Med. 2022 Nov 20;11(22):6848. doi: 10.3390/jcm11226848. PMID 36431325
- [Background] Tritos NA, Biller BMK. Current management of Cushing's disease. J Intern Med. 2019 Nov;286(5):526-541. doi: 10.1111/joim.12975. Epub 2019 Oct 4. PMID 31512305
- [Background] Pivonello R, De Martino MC, De Leo M, Simeoli C, Colao A. Cushing's disease: the burden of illness. Endocrine. 2017 Apr;56(1):10-18. doi: 10.1007/s12020-016-0984-8. Epub 2016 May 17. PMID 27189147
- [Background] Pecori Giraldi F, Moro M, Cavagnini F; Study Group on the Hypothalamo-Pituitary-Adrenal Axis of the Italian Society of Endocrinology. Gender-related differences in the presentation and course of Cushing's disease. J Clin Endocrinol Metab. 2003 Apr;88(4):1554-8. doi: 10.1210/jc.2002-021518. PMID 12679438
- [Background] Nishioka H, Yamada S. Cushing's Disease. J Clin Med. 2019 Nov 12;8(11):1951. doi: 10.3390/jcm8111951. PMID 31726770